CLINICAL TRIAL: NCT05984901
Title: Continuous Ambulatory Vestibular Assessment (CAVA): Development of a System to Provide an Automatic Diagnosis for Vestibular Conditions
Brief Title: The CAVA Multicentre Dizziness Trial
Acronym: CAVA 2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Norfolk and Norwich University Hospitals NHS Foundation Trust (Other)
Collaborators: University Hospitals, Leicester (Other); St George's University Hospitals NHS Foundation Trust (Other); Gloucestershire Hospitals NHS Foundation Trust (Other); University Hospital Birmingham NHS Foundation Trust (Other); Mid and South Essex NHS Foundation Trust (Other); Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRAS: 317899
Record Dates: First submitted 2023-05-02; First posted 2023-08-09 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-03

CONDITIONS: Ménière's Disease; Vestibular Migraine; Benign Paroxysmal Positional Vertigo (BPPV)
MeSH Terms: conditions — Meniere Disease; Benign Paroxysmal Positional Vertigo | interventions — Drug Delivery Systems

STUDY DESIGN:
Intervention Model Description: All participants fulfilling the eligibility criteria and providing consent will wear the CAVA device for 30 days. The CAVA algorithm will then diagnose each patient based only on the data recorded from the device. The accuracy of the system will be tested by comparing the CAVA system's diagnosis with each patient's known diagnosis. The results of the algorithm work ("the diagnosis") will not be available until the end of the trial and will not be made available to clinicians or patients during the trial.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The CAVA Multicentre Dizziness Trial (CAVA2) (Other): CAVA 2 is a single arm study testing a diagnostic device to diagnose different inner-ear conditions appraised by calculating values for sensitivity and specificity. Head and eye movements recorded by the CAVA device will enable the computer algorithms (to be developed) to differentiate between the three target conditions.
  Interventions: Device: The continuous ambulatory vestibular assessment (CAVA) system

INTERVENTIONS:
Device: The continuous ambulatory vestibular assessment (CAVA) system — The CAVA trial is a diagnostic accuracy multicentre device trial which aims to quantify the extent to which the CAVA system can differentiate three common inner-ear causes of dizziness: Ménière's disease, vestibular migraine and Benign Paroxysmal Positional Vertigo (BPPV).
  The CAVA device is composed of two components: a set of bespoke single-use sensor arrays that adhere to the left and right side of the participant's face; and a small reusable module fitting over the ear that contains a battery, microcomputer data storage facility and connection ports for the arrays. The CAVA device will be worn by all participants for 30 days with the aim of capturing eye movement data during a dizzy attack.
  The first objective is to develop an algorithm that can discriminate between the 3 listed dizziness conditions. The second is to quantify the financial and patient benefits of deployment in the NHS. The final objective is to expedite a plan to deploy the system in the NHS.

SUMMARY:
The CAVA trial is a diagnostic accuracy multicentre device trial which aims to quantify the extent to which the CAVA system can differentiate three common inner-ear causes of dizziness: Ménière's disease, vestibular migraine and Benign Paroxysmal Positional Vertigo (BPPV).

The CAVA device is composed of two components: a set of bespoke single-use sensor arrays that adhere to the left and right side of the participant's face; and a small reusable module fitting over the ear that contains a battery, microcomputer data storage facility and connection ports for the arrays. The CAVA device will be worn by all participants for 30 days with the aim of capturing eye movement data during a dizzy attack.

The first objective is to develop an algorithm that can discriminate between the 3 listed dizziness conditions. The second is to quantify the financial and patient benefits of deployment in the NHS. The final objective is to expedite a plan to deploy the system in the NHS.

DETAILED DESCRIPTION:
This is a multicentre diagnostic accuracy study with a recruitment target of 255 adult participants. Recruitment will take place across ten sites in the UK, over two years. To be eligible, participants must have an existing diagnosis of Ménière's disease, vestibular migraine or BPPV. The study will recruit eighty-five participants with each condition. Each patient's diagnosis will form the "reference standard" which will later be compared with a automated computer diagnosis.

Each participant will wear the CAVA device near continuously for thirty days. The device will record all eye and head movements during this time, including during any episodes of vertigo. When a patient experiences an episode of vertigo, they will be asked to activate an event marker on the CAVA device and keep a written record of attack onset and duration in a diary. Although this manual logging will not be relied upon for algorithm development, the whole 30 days of data will be used to detect periods of eye movement associated with dizziness.

The investigators will develop computer algorithms that use the data captured by the CAVA devices to differentiate between three target conditions. These algorithms will build on the algorithms that have been developed during the current MRC grant which have produced excellent results.10,11,17. The algorithms use deep learning neural networks (DNNs) in a so-called 'end-to-end' approach. In this approach, a multi-layered network takes as input 'raw' time domain data and outputs a classification decision without using any explicit intermediate representations of the signal (such as signal entropy, power, skewness, kurtosis etc.). End-to-end approaches, which typically utilise alternating sequences of convolution and pooling layers, fully connected layers, auto-encoders and long short-term memory (LSTM) layers, have been shown to outperform traditional approaches in cases where large amounts of training data are available. However, they provide little insight into how they work (i.e., which features of the signal are important for classification). It will therefore also be considered to develop methods in which intermediate representations are generated and then use these input features to test a range of classifiers (e.g., boosted trees, random forests, logistic regression, support vector machines etc.).

The performance of the algorithms will be assessed using the 'leave-one-out cross-validation' technique, which is the usual way of evaluating classifiers.22 In this technique, the data from a single patient is set aside and the remaining data from the other patients is used to 'train' the classifier. A algorithm will be referred to that is trained to distinguish the three conditions as a 'classifier'. The classifier is then tested on the set aside data: the testing process consists of comparing the classifier's predicted diagnosis ('Ménière's disease', 'vestibular migraine' or 'BPPV') with the true diagnosis (the reference standard label). This process is repeated, removing a different patient's data each time, producing an automated diagnosis for all 255 patients. Although computationally expensive, this ensures that the classifier has not 'seen' during training the data from the patient it tests, which would bias its decision. It also closely matches the real-world scenario of a new patient presenting to their clinician and a diagnosis being provided on the basis of their experience of other patients.

The study will present the sensitivity and specificity for diagnosing each of the three target conditions and Receiver Operator Curves (ROCs), showing how the diagnostic accuracy changes for various classification thresholds.

The target conditions have different incidences. Reflecting this imbalance in this study's statistical calculations would require many thousands of patients with the most common of these conditions. It is believed that this would not be economically viable and would not add value to the study. The results obtained will be sufficiently robust to demonstrate the system's efficacy and the expected detection rate for each disease.

A Health Economist (HE) will assess the potential resource, financial savings and patient benefits of a diagnostic pathway incorporating CAVA compared to existing pathways. The study design ensures that appropriate data collection is embedded into the study for the economic evaluation. An early cost-effectiveness model will be developed using retrospective patient data (e.g., history, number of tests and hospital visits). The model will reveal the potential savings and benefits of CAVA's predictive algorithms at various hypothetical thresholds of diagnostic accuracy versus a standard diagnostic pathway. A counterfactual pathway of diagnosis with the CAVA device will be developed against standard of usual care at the moment, to inform the most likely potential economic benefits.

A commercialisation consultant will oversee a portfolio of work to support the commercialisation of the CAVA system. They will produce a market access plan detailing CAVA's route to commercialisation and confirm CAVA's placement within existing NHS pathways and how it would be implemented. The Investigators will build upon the previous focus-group work with a stakeholders' event involving professionals, patients, and IT stakeholders from NHS organisations. The investigators will identify the issues important to stakeholders regarding the feasibility of adoption within the NHS and will establish support for adoption. A PPI event will be hosted to review the interim findings from the trial and a public dissemination event to share the findings with the public. Throughout the project prospective licenses will be engaged.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 and over
2. Must have relevant index medical condition: Ménière's Disease, Vestibular Migraine, posterior canal Benign Paroxysmal Positional Vertigo (see section 6.3.1.2 for specific criteria)
3. Experiencing episodes of true vertigo with at least 2 episodes within the preceding 4 weeks at time of consent
4. The duration and nature of the vertigo is of a duration and a nature supportive of the relevant index medical condition
5. Owns and able to use a telephone
6. Willing to provide informed consent
7. Willing to comply with the study protocol for using the CAVA device
8. Willing to complete all study materials
9. Adequate grasp of the English language or language used within an existing translated version of the informed consent form and patient information sheet and where hospital translators are available to provide support

Exclusion Criteria:

1. Has an allergy to plasters and/or medical adhesives
2. Evidence of dermatitis, fragile skin, or any other condition that could be aggravated by the repeated application of skin surface adhesives
3. Pregnant or breastfeeding mothers
4. Bilateral or second side Ménière's Disease
5. Active bilateral or second side posterior canal Benign Paroxysmal Positional Vertigo
6. Currently enrolled on an intervention trial (not including questionnaire-based or observational trial)
7. Patients who meet diagnostic criteria for more than one eligible condition at time of recruitment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Success of a diagnostic device to diagnose different inner-ear conditions | 30 Days
  The primary outcome is the success of a diagnostic device to diagnose different inner-ear conditions appraised by calculating values for sensitivity and specificity. Head and eye movements recorded by the CAVA device will enable the computer algorithms (to be developed) to differentiate between the three target conditions.
  The investigators will develop computer algorithms that use the data captured by the CAVA devices to differentiate between the three target conditions. The algorithms use deep learning neural networks (DNNs) in a so-called 'end-to-end' approach. In this approach, a multi-layered network takes as input 'raw' time domain data and outputs a classification decision without using any explicit intermediate representations of the signal (such as signal entropy, power, skewness, kurtosis etc.)

SECONDARY OUTCOMES:
Health economics data | 30 Days
  Health economics data will inform analysis of potential financial and patient benefits of a diagnostic pathway incorporating the CAVA system compared to existing pathways. An early cost-effectiveness model will be developed using retrospective patient data.
  The data will be used to estimate the frequency of likely NHS resource-use of patients under observation with one of the three diagnoses, to determine the likely cost and Health-related quality of life impacts of each. It will also be used to assess the prevalence of time-off-work (productivity), reduced productivity and reduce non-paid activities e.g., volunteering, caring etc. as well as insights into early- retirements or changes in occupation etc.

CONTACTS AND LOCATIONS:
Overall Officials: John Phillips, PhD, Principal Investigator — Consultant ENT Surgeon
Locations (1):
- Norfolk and Norwich University Hospitals Foundation Trust, Norwich, Norfolk, United Kingdom